CLINICAL TRIAL: NCT04867733
Title: Evaluating Racial and Ethnic Differences in Dermal Micropore Formation Using Optical Coherence Tomography
Brief Title: Visualizing Dermal Micropores With OCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Nicole K Brogden, Associate Professor, University of Iowa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2020010229
Record Dates: First submitted 2021-04-29; First posted 2021-04-30 (Actual); Results first posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2023-12

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Micropatch application (Experimental): All participants will complete this arm. Three sites each on the upper arm, volar (inner) forearm, and palm will be identified. Baseline measurements of trans-epidermal water loss, electrical resistance, and color will be made at each site. Baseline optical coherence tomography (OCT) scans will be made at each site. Color will only be measured at baseline. One site at each location will undergo the following interventions: 1) micropatch application and an occlusive covering, 2) micropatch application, but remain uncovered, 3) occlusive covering, no micropatch application. Micropatch application will only occur on the first day and does not contain any drug substance. Trans-epidermal water loss and electrical resistance are re-measured after micropatch removal, along with an additional OCT scan. Electrical resistance and OCT scans will be repeated at all sites for 2 days. Measurements from the 2nd and 3rd sites allow each subject to serve as their own control in data analysis.
  Interventions: Other: Micropatch (microneedle patch)

INTERVENTIONS:
Other: Micropatch (microneedle patch) — Each micropatch contains an array of 50 microneedles.

SUMMARY:
The study to be performed will allow visualization of skin micropores following microneedle treatment in healthy subjects in differing racial/ethnic backgrounds.

DETAILED DESCRIPTION:
Transdermal drug delivery (by way of patches that adhere to the skin and deliver drug in a time-dependent fashion) allows for systemic drug delivery through the skin, while avoiding many of the side effects and challenges associated with oral or intravenous drug delivery. One significant challenge limiting the number of drug compounds that can be transdermally delivered is the hydrophobic nature of the skin, which provides a highly efficient barrier against the absorption of drug molecules. Micropatches are small patches with tiny projections that are a minimally invasive way to allow drug molecules to cross the skin by creating micron-sized channels (also called micropores) in the skin, thereby increasing its permeability. Micropatches have been safely used in hundreds of patients for administration of drugs and vaccines through the skin. Studies have demonstrated that micropatch treatment is relatively painless and well-tolerated by most patients.

Following micropatch treatment, the skin must heal the micropores. In young healthy individuals this process takes approximately 48 to 72 hours when the skin is covered by an occlusive patch. One of the factors that may also affect micropore healing time is the depth of the micropores in the skin immediately after micropatch treatment. There are almost no data available regarding how race and ethnicity affect the depth of micropores after micropatch application. It is important to study differences in micropore depth so investigators can better understand why rates of micropore closure vary in different racial/ethnic populations. Without this information the potential for variability in drug delivery is high.

In this study the investigators will objectively measure skin color with a colorimeter to characterize the epidermal properties of individuals of different self-identified races and ethnicities. Measurements of trans-epidermal water loss will be used to evaluate formation of micropores in the skin; electrical impedance measurements will be used to estimate rates of micropore closure. The investigators will visualize the micropores created after micropatch treatment with the use of an optical coherence tomography instrument that will allow for calculation of epidermal thickness and micropore depth. All of these skin characteristics can be measured using noninvasive methods that are quick and painless.

ELIGIBILITY:
Inclusion Criteria: Subjects will be healthy men and women between 18 and 45 years of age.

Exclusion Criteria:

1. Unable to give consent
2. Severe general allergies requiring chronic treatment with steroid or antihistamines
3. Previous adverse reaction to microneedle insertion
4. History of keloids
5. Known allergy or adverse reaction to medical tape/adhesive, or aloe vera
6. Any inflammatory diseases of the skin (including but not limited to: psoriasis, atopic dermatitis, and blistering skin disorders)
7. Any disease associated with altered immune function (including but not limited to: rheumatoid arthritis, diabetes, lupus, HIV/AIDS)
8. Any subject taking medication that impairs the immune system (including but not limited to corticosteroids, TNF inhibitors, monoclonal antibodies, chemotherapy agents)
9. Any current malignancy or history of malignancy present at the treatment sites
10. Eczema or scaling present at any treatment site; any current inflammation or irritation present at the treatment sites (including but not limited to: rash, inflammation, erythema, edema, blisters)
11. Uncontrolled mental illness that would, in the opinion of the investigator, affect the subject's ability to understand or reliably participate in the study
12. Subjects taking medications in the following therapeutic classes will be excluded: HMGCoA reductase inhibitors ("statins"), oral or topical steroids (at the local treatment site), oral antibiotics, topical antibiotics at the local treatment site, topical antihistamines at the local treatment site, beta-blockers, and systemic or topical NSAIDS/analgesics. A subject who has recently used oral or topical steroids, antibiotics, antihistamines, or analgesics may be enrolled if more than 5 elimination half-lives of the drug have passed since the last dose (this is a typical parameter in pharmacokinetics, when it is assumed that ~97% of drug in the systemic circulation is eliminated after 5 half-lives). The estimated elimination half-life for any specific drug will be obtained from standard pharmacy references such as Micromedex or other comparable drug information references.
13. Any subjects that are pregnant/nursing will be excluded from participation.
14. Subjects will also be excluded for any condition that would, in the opinion of the PI or physician, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-06-29 (Actual); Study Completion 2022-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Brogden, PharmD, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cota V, Brogden NK. Micropore visualization and lifetime following microneedle application to skin of differing pigments. Drug Deliv Transl Res. 2025 Oct;15(10):3528-3541. doi: 10.1007/s13346-025-01817-9. Epub 2025 Mar 5. PMID 40042738

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Micropatch Application
Started | 49
Completed | 49
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Micropatch Application
Number analyzed (Participants) | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 44
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 13
  More than one race | 14
  Unknown or Not Reported | 5

OUTCOME MEASURES:

1. Primary Outcome: Micropore Depth, Upper Arm
Description: The depth of the micropore created at the upper arm will be measured using OCT scans. These data are only collected from the micropatch sites. Data will be calculated as the mean of micropore depth measured at all micropatch sites.
Time Frame: Post microneedle application (Day 0), approximately 5 minutes
Measure: Mean (Standard Deviation); unit: micrometer
Arm/Group | Micropatch Application
Number analyzed (Participants) | 49
micrometer | 72.4 (10.7)

2. Primary Outcome: Micropore Depth, Volar Forearm
Description: The depth of the micropore created at the volar forearm will be measured using OCT scans. These data are only collected from the micropatch sites. Data will be calculated as the mean of micropore depth measured at all micropatch sites.
Time Frame: Post microneedle application (Day 0), approximately 5 minutes
Measure: Mean (Standard Deviation); unit: micrometer
Arm/Group | Micropatch Application
Number analyzed (Participants) | 49
micrometer | 78.6 (12.6)

3. Primary Outcome: Micropore Depth, Palm
Description: The depth of the micropore created at the palm will be measured using OCT scans. These data are only collected from the micropatch sites. Data will be calculated as the mean of micropore depth measured at all micropatch sites.
Time Frame: Post microneedle application (Day 0), approximately 5 minutes
Measure: Mean (Standard Deviation); unit: micrometer
Arm/Group | Micropatch Application
Number analyzed (Participants) | 49
micrometer | 102.8 (21.2)

4. Secondary Outcome: Change in Trans-epidermal Water Loss, Upper Arm
Description: The percent change in trans-epidermal water loss from baseline to post-micropatch application at the upper arm sites will be calculated. These data are only collected from the micropatch sites. Percent change is calculated as (trans-epidermal water loss after micropatch application/baseline trans-epidermal water loss) x 100. Data will be calculated as the mean of measurements from the micropatch sites at the upper arm.
Time Frame: Baseline (Day 0) and post-microneedle application (Day 0), approximately 1-3 minutes
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Micropatch Application
Number analyzed (Participants) | 49
percentage change from baseline | 267.4 (95.8)

5. Secondary Outcome: Change in Trans-epidermal Water Loss, Volar Forearm
Description: The percent change in trans-epidermal water loss from baseline to post-micropatch application at the volar forearm sites will be calculated. These data are only collected from the micropatch sites. Percent change is calculated as (trans-epidermal water loss after micropatch application/baseline trans-epidermal water loss) x 100. Data will be calculated as the mean of measurements from the micropatch sites at the volar forearm.
Time Frame: Baseline (Day 0) and post-microneedle application (Day 0), approximately 1-3 minutes
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Micropatch Application
Number analyzed (Participants) | 49
percentage change from baseline | 313.2 (112.3)

6. Secondary Outcome: Change in Trans-epidermal Water Loss, Palm
Description: The percent change in trans-epidermal water loss from baseline to post-micropatch application at the palm sites will be calculated. These data are only collected from the micropatch sites. Percent change is calculated as (trans-epidermal water loss after micropatch application/baseline trans-epidermal water loss) x 100. Data will be calculated as the mean of measurements from the micropatch sites at the palm.
Time Frame: Baseline (Day 0) and post-microneedle application (Day 0), approximately 1-3 minutes
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Micropatch Application
Number analyzed (Participants) | 49
percentage change from baseline | 131.3 (46.1)

7. Secondary Outcome: Skin Color
Description: Lightness/darkness of the skin color is measured with a tristimulus colorimeter and reported in a unitless scale called the CIELAB color space (sometimes also called the L*a*b* color space). In this study we measured the value called L*. The L* values can range from 0 (black) to 100 (white). Higher L* values denote lighter skin, while lower L* values denote darker skin. The L* measurement is an objective measurement of skin color and there is no "better" or "worse" values of L*. The L* values are collected from the all 9 sites (3 each at upper arm, volar forearm, and palm) and the measurements are averaged together and reported as the mean.
Time Frame: Baseline (Day 0), <30 seconds
Measure: Mean (Standard Deviation); unit: L* (unitless measure on a scale)
Arm/Group | Micropatch Application
Number analyzed (Participants) | 49
L* (unitless measure on a scale) | 58.9 (8.6)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored during the 3 days while a subject was completing the study and for three days after study completion.
Arm/Group | Micropatch Application
All-Cause Mortality (participants affected / at risk) | 0/49
Serious Adverse Events (participants affected / at risk) | 0/49
Other Adverse Events (participants affected / at risk) | 3/49
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Micropatch Application (N=49)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-12): https://cdn.clinicaltrials.gov/large-docs/33/NCT04867733/Prot_SAP_000.pdf